CLINICAL TRIAL: NCT02236208
Title: Mechanism of Folate Acid in Influencing Offspring Obesity During Pregnancy
Brief Title: Effect of Folate Acid on Offspring Obesity
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xirong Guo, Vice-president of Nanjing Maternity and Child Health Care Hospital, Nanjing Medical University
Other Study IDs: NMU-530604-XG1
Record Dates: First submitted 2014-09-02; First posted 2014-09-10 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to observe the effect of lack or excess of folic acid in first, second and third trimester on child birth weight, fat content and the secretion of metabolism related hormone, and clinical follow-up their offspring obesity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy women
* children
* Chinese

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with the early, mid and late pregnancy; Chilren
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
The level of folate acid of pregnancy women at first trimester | 12 weeks of pregnancy

SECONDARY OUTCOMES:
The level of folate acid of pregnancy women at second trimester | 20-24 weeks of pregnancy
The level of folate acid of pregnancy women at third trimester | 28-40 weeks of pregnancy
The birth weight, fat content and metabolism related hormone secretion of their offspring | At birth
The weight, fat content and metabolism related hormone secretion of their offspring at one year old | One years old
The weight, fat content and metabolism related hormone secretion of their offspring at 3 years old | 3 years old
The weight, fat content and metabolism related hormone secretion of their offspring at 5-7 years old | 5-7 years old
The weight, fat content and the secretion of metabolism related hormone of offspring at 18 years old | 18 years old

CONTACTS AND LOCATIONS:
Overall Officials: Xirong Guo, Dr., Principal Investigator — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China